CLINICAL TRIAL: NCT05469503
Title: A Randomized, Placebo-controlled, Double-blind Study to Assess the Effect of TOTUM-854 on Blood Pressure in Subjects With Moderately Elevated Blood Pressure
Brief Title: Effect of TOTUM-854 on Blood Pressure in Subjects With Moderately Elevated Blood Pressure
Acronym: INSIGHT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: Excelya (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VCT-009; 2022-A00131-42 (Other: ID-RCB)
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Prehypertension; Elevated Blood Pressure; Blood Pressure; Metabolic Syndrome
Keywords: Diet supplement; Plant extracts; Hygiene and dietary recommendations
MeSH Terms: conditions — Prehypertension; Hypertension; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOTUM-854 (Experimental): Experimental active diet supplement TOTUM-854 3.71-g dose. Seven capsules per day to consume orally in two intakes
  Interventions: Dietary Supplement: TOTUM-854
- Placebo (Placebo Comparator): Placebo comparator Seven capsules per day to consume orally in two intakes
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: TOTUM-854 — 12 weeks of TOTUM-854 supplementation
  Arms: TOTUM-854
Dietary Supplement: Placebo — 12 weeks of placebo supplementation
  Arms: Placebo

SUMMARY:
This clinical study aims to assess the efficacy of TOTUM-854, a mix of 6 plant extracts, consumed twice a day on automated office blood pressure in subjects with moderately elevated blood pressure. The hypothesis is that TOTUM-854 is superior to placebo for decrease of automated office blood pressure after 12 weeks of consumption.

ELIGIBILITY:
Main Inclusion Criteria:

* Office Systolic Blood Pressure between 130 and 159 mmHg and Diastolic Blood Pressure < 100 mmHg
* Body Mass Index (BMI) between 18.5 and 35 kg/m²
* Weight stable within ± 5 % in the last three months
* No significant change in food habits or in physical activity in the 3 months before the randomization and agreeing to keep them unchanged throughout the study

Main Exclusion Criteria:

* Known or suspected secondary hypertension
* Subjects with a very high Cardio Vascular risk SCORE2 or SCORE2-OP according to their risk regions: (Subjects <50 years old: ≥7.5%; Subjects between 50 and 69 years old: ≥10%; Subjects ≥70 years old: ≥15%)
* Known hypertensive retinopathy and/or hypertensive encephalopathy
* History of spontaneous or drug-induced angioedema
* Clinically significant valvular heart disease or severe aortic stenosis
* History of an acute coronary syndrome (non-ST elevation myocardial infarction, ST-elevation myocardial infarction, and unstable angina pectoris), stroke, or transient ischemic attack within 6 months prior to inclusion
* Newly diagnosed or suffering from a non-treated or uncontrolled metabolic disorder such as diabetes, dyslipidemia, thyroidal dysfunction or other metabolic disorder
* Suffering from a severe chronic disease or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure at V4 | V4 (12 weeks of intervention)
  Automated Office Blood Pressure (in mmHg), TOTUM-854 vs placebo

SECONDARY OUTCOMES:
Evolution of Systolic Blood Pressure | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks) and V5 (4 weeks after the stop of intervention)
  Automated Office Blood Pressure (in mmHg), TOTUM-854 vs placebo
Evolution of Diastolic Blood Pressure | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  Automated Office Blood Pressure (in mmHg), TOTUM-854 vs placebo
Evolution of the fasting blood glycemia | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  Glycemia (in mg/dL), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of triglycerides | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  Triglycerides (in g/L), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of total cholesterol | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  Total cholesterol (in g/L), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of HDL cholesterol | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  HDL cholesterol (in g/L), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of non-HDL cholesterol | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  non-HDL cholesterol (in g/L), TOTUM-854 vs placebo
Evolution of the fasting blood concentration of LDL cholesterol (Friedewald method) | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  LDL cholesterol (in g/L, Friedewald method), TOTUM-854 vs placebo
Evolution of the fasting blood hsCRP concentration | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  hsCRP (in mg/L), TOTUM-854 vs placebo
Evolution of the body weight | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  Body weight (in kg), TOTUM-854 vs placebo
Evolution of the waist circumference | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  Waist circumference (in cm), TOTUM-854 vs placebo
Evolution of the hip circumference | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  Hip circumference (in cm), TOTUM-854 vs placebo
Evolution of the cardiovascular disease risk (SCORE value) | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  Systematic Coronary Risk Estimation value from Heartscore calculator, TOTUM-854 vs placebo
Delay of occurence of pharmacological treatment requirement for hypertension from V1 | V1 (baseline), V2 (4 weeks of intervention), V3 (8 weeks), V4 (12 weeks) and V5 (4 weeks after the stop of intervention)
  Delay between V1 and the date at which the investigator will decide to withdraw the subject from the study because he needs a pharmacological treatment to treat his hypertension, TOTUM-854 vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Pałka, Dr, Principal Investigator — Centrum Medyczne Linden
Locations (10):
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment Cardiology Department, Haskovo
  - Multiprofile Hospital for Active Treatment - Uni Hospital OOD, Cardiology Department, Panagyurishte
  - Diagnostic Consultative Center VII-Plovdiv South district EOOD, Cabinet of Endocrinology, Plovdiv
  - Multiprofile Hospital for Active Treatment Sveta Karidad EAD, Cardiology Department, Plovdiv
  - Diagnostic Consultative Center XX- Sofia EOOD, Sofia
- CHU Clermont Ferrand PIC/CIC Inserm 1405, Clermont-Ferrand, France
- Poland (4):
  - Vitamed Gałaj i Cichomski sp.j, Bydgoszcz
  - Centrum Medyczne Linden, Krakow
  - Przychodnia Zespołu Lekarza Rodzinnego "Medyk", Słupca
  - Centrum Medyczne Oporów, Wroclaw